CLINICAL TRIAL: NCT04514029
Title: Neurotoxicity Prophylaxis With Intrathecal Dexamethasone and Simvastatin in Adults Receiving Axicabtagene Ciloleucel (Axi-Cel) Treatment
Brief Title: Neurotoxicity Prophylaxis With Intrathecal Dexamethasone and Simvastatin Post Axi-Cel
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019LS161
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
Keywords: Lymphoma; CAR-T; Neurotoxicity; CRS; Dexamethasone; Simvastatin
MeSH Terms: conditions — Lymphoma; Neurotoxicity Syndromes | interventions — Simvastatin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Simvastatin and Dexamethasone (Experimental): Simvastatin 40 mg/day will be started at least 5 days prior to apheresis and will be continued until day +30 after infusion. Intrathecal dexamethasone 8 mg will be administered on days (related to CAR-T infusion) -1, +6, +13, (+/- 2 days).
  Interventions: Drug: Simvastatin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg started 2 weeks (+/-5 days) prior to apheresis through day +30
Drug: Dexamethasone — Intrathecal dexamethasone 8 mg on days -1, +6, +13 (+/-2 days)

SUMMARY:
Open-label, single-arm, single center pilot study to assess safety and feasibility of administering dexamethasone intrathecally and simvastatin orally during axicabtagene ciloleucel (axi-cel) treatment. Feasibility will be measured by the proportion of patients completing two-thirds (2/3) of their assigned treatments. The study will be deemed feasible if 2/3 or more of the patients complete 2/3 or more of their allocated treatments.

DETAILED DESCRIPTION:
This trial gathers preliminary information on the potential effect of the combination of dexamethasone and simvastatin on treating Neurotoxicity (NT) in the patient population. The rate of patients completing all required study treatments and the rate of NT will be determined.

Simvastatin 40 mg/day will be started at least 5 days prior to apheresis and will be continued until day +30 after infusion. Intrathecal dexamethasone 8 mg will be administered on days (related to CAR-T infusion) -1, +6, +13, (+/- 2 days). CSF samples (3 ml) will be collected at these time points. Peripheral blood samples of 4 ml will be collected on days -1, +1, +6, and +13. The care team will check weekly CK and LFTs to ensure safety of simvastatin. Patients who develop NT will be allowed to continue treatment if feasible along with standard of care management.

ELIGIBILITY:
Inclusion Criteria:

* 18- 80 years of age
* One of the following histologies:

  * Diffuse large B-cell lymphoma (DLBCL) not otherwise specified, or
  * Primary mediastinal B-cell lymphoma, or
  * High grade B-cell lymphoma, or
  * DLBCL arising from follicular lymphoma
* Disease status:

  * Chemotherapy refractory disease after ≥2 lines of chemotherapy, or
  * Relapsed with no remission after ≥1 lines of salvage chemotherapy, or
  * Relapsed following autologous hematopoeitic stem cell transplantation (and failed at least 2 prior lines of therapy including high dose chemotherapy). If salvage therapy is given post auto HCT, the subject must have no complete response, or relapse after the last line of therapy
* Performance Status

  * ECOG performance status 0-2
* Adequate organ function defined as:

  * Renal function defined as:

    * eGFR ≥ 30 mL/min/1.73 m^2
  * Liver function defined as:

    * ALT and AST ≤ 5 times the ULN for age (unless due to disease)
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
  * Hemodynamically stable and LVEF ≥ 40% confirmed by echocardiogram or MUGA
* Women of childbearing potential and men with partners of child-bearing potential must agree to use of contraception for the duration of treatment as outlined in axi-cel protocol.
* Able to provide written voluntary consent (or LAR consent for adults with diminished capacity) prior to the performance of any research related tests or procedures
* Availability of a certified practitioner to perform the lumbar punctures

Exclusion Criteria:

* Allergies, or intolerance to simvastatin or dexamethasone
* Already receiving a statin drug for hypercholesterolemia and unwilling to change medication to 40 mg/day of simvastatin
* Active uncontrolled CNS lymphoma. Patients with history of CNS lymphoma who have been adequately treated are eligible
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD).
* Uncontrolled active hepatitis B or hepatitis C
* Active HIV infection
* Uncontrolled acute life threatening bacterial, viral or fungal infection
* Unstable angina and/or myocardial infarction
* Risk factors that preclude a safe lumbar puncture (high intracranial pressure, bleeding diathesis that cannot be reversed or corrected, need for uninterrupted anticoagulation, platelets < 50K that cannot be corrected with transfusional support
* Pregnant or breastfeeding as agents used in this study are Pregnancy Category C (dexamethasone) and X (simvastatin). Females of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days of study registration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients completing two-thirds of their assigned treatment | 30 days after initiation of CAR-T therapy
  The feasibility of administering Simvastatin and Dexamethasone will be measured by the proportion of the patients completing two-thirds (2/3) of their assigned treatments.
Number of patients experiencing adverse events | From the day of 1st dose of simvastatin and until day +7 after the last dose of simvastatin.
  Safety of administering Simvastatin and Dexamethasone will be measured by the proportion of patients experiencing adverse events related to the study treatment.

SECONDARY OUTCOMES:
The change in IL-6 levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
The change in IL-8 levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
The change in IL-10 levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
The change in MCP-1 levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
The change in VEGF levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
The change in PDGFR levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
The change in cleaved-caspase 3 levels | One day prior to infusion and at days +1,+6, and +13 post infusion
  Pre- and post-infusion levels of a cytokine profile will be measured by a Lumina multiplex array in the serum and CSF of patients at time of CRS and NT if samples available.
Number of participants experiencing severe NT | 30 days after initiation of CAR-T therapy
  The incidence of severe NT in patients receiving CAR-T cell dexamethasone and simvastatin.
Number of participants experiencing overall best response with CAR-T cell therapy | 30 days after initiation of CAR-T therapy
  The overall response rate of CAR-T cells as defined by Lugano criteria.
The change in serum levels of ANG1 with statin therapy | 30 days after initiation of CAR-T therapy
  ANG1 levels in serum will be measured using an enzyme-linked immunosorbent assay (ELISA)
The change in serum levels of ANG2 with statin therapy | 30 days after initiation of CAR-T therapy
  ANG2 levels in serum will be measured using an enzyme-linked immunosorbent assay (ELISA)
The change in serum levels of IP10 with statin therapy | 30 days after initiation of CAR-T therapy
  IP10 levels in serum will be measured using an enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Maakaron, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States